CLINICAL TRIAL: NCT06898333
Title: Evaluating the Implementation and Effectiveness of the BJC-Pink and Pearl Project on Lung Cancer Screening
Brief Title: Implementation and Effectiveness of the BJC-Pink and Pearl Project on Lung Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202412064
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; Cancer of the Lung
Keywords: Lung cancer screening (LCS); Pink and Pearl Campaign; Breast cancer screening (BCS); Low-dose computed tomography (LDCT); Smoking history; Health disparities; Screening behavior; Feasibility; Acceptability; Appropriateness
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants - scheduled for mammography and eligible for LCS: Women who are scheduled for mammography and are potentially LCS-eligible will be approached by the registration team and will complete a survey. Subjects who were referred for LCS will be contacted and the investigators will gauge their interest in returning for dual breast and lung screening program in future and rate their experience on a patient satisfaction scale.
- Providers: Providers in the breast radiology service who referred women to LCS. Investigators will gather information on the feasibility, acceptability, and appropriateness of the Pink and Pearl project.

SUMMARY:
The investigators proposal is ripe for executing as the investigators seek to leverage this "natural experiment" initiated by the BJC health system to evaluate the effectiveness of the Pink & Pearl Campaign as an implementation strategy to promote lung cancer screening (LCS) uptake among LCS-eligible women undergoing mammography at BJC West County. This evaluation is grounded in the Integrated Screening Action Model that depicts individual- and environmental-level influences on the screening behavior process. Using an explanatory sequential mixed methods design, which combines both quantitative and qualitative approaches, the research questions and specific aims for this proposal are to: a) evaluate the baseline prevalence of LCS among LCS-eligible women; b) assess whether the Pink & Pearl Campaign increases referrals and uptake/ completion of LCS among LCS-eligible women undergoing screening mammography; and c) evaluate individual and environmental factors influencing LCS uptake, and implementation outcomes of the campaign. These implementation outcomes will help identify whether the campaign was put in place successfully or not. This proposal will inform strategies for integrating cancer screening programs to improve poorly performing programs like LCS.

ELIGIBILITY:
Inclusion Criteria for Participants:

* Undergoing screening mammography
* Between the ages of 50-80 years (inclusive)
* Reporting a 20 pack-year equivalent of either current smoking history or have quit in the past 15 years
* Can speak and understand English
* Ability to understand willingness to provide informed consent.

Exclusion Criteria for Participants:

* Diagnosed with a serious health problem that will likely limit life expectancy (such as previous history of lung cancer, symptoms of lung cancer such as hemoptysis or unexplained weight loss of more than 6.8 kg (15 lb) in the previous year)

  * Subjects with symptoms of lung cancer should get a diagnostic CT scan
* Unable or unwilling to get treatment if lung cancer is found

Eligibility Criteria for Providers:

* Older than 20 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women within the BJC West County electronic health record (EHR) who are scheduled to undergo screening mammography and are eligible for LCS, based on 2021 USPSTF guidelines. In addition to patients, healthcare providers involved in the breast radiology service who referred women to the Pink and Pearl project will also be included as study participants for the qualitative in-depth interviews. This group may include medical doctors, nurse practitioners, nurses, nurse navigators, and physician assistants. Up to 15 healthcare providers will be interviewed.
Sampling Method: Non-Probability Sample
Enrollment: 279 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of LCS-eligible women who opt-in to, and successfully, complete LCS mammography and opt-in to lung cancer screening | At baseline
Number of women screened for LCS | At 3 months
Number of women screened for LCS | At 6 months
Feasibility of Pink and Pearl project | At 6 months
  Feasibility is defined as the extent to which the strategy is suitable for routine use in a setting.
  Information on the feasibility of the Pink and Pearl campaign from healthcare providers will be collected using in-depth interviewing.
Acceptability of Pink and Pearl project | At 6 months
  Acceptability is defined as the perception that the strategy is agreeable or satisfactory.
  Information on the acceptability of the Pink and Pearl campaign from healthcare providers will be collected using in-depth interviewing.
Appropriateness of Pink and Pearl project | At 6 months
  Appropriateness is defined as the perceived fit, relevance, or compatibility of the strategy or practice for a given setting.
  Information on the appropriateness of the Pink and Pearl campaign from healthcare providers will be collected using in-depth interviewing.

SECONDARY OUTCOMES:
Median time to lung cancer screening | Through completion of follow-up (estimated to be 1 year)
Number of women who have a positive lung radiology screening | Through completion of follow-up (estimated to be 1 year)
Rate of follow-up for a positive screening examination | Through completion of follow-up (estimated to be 1 year)
False positive rates | Through completion of follow-up (estimated to be 1 year)
Invasive intervention rate | Through completion of follow-up (estimated to be 1 year)
  Invasive interventions are considered percutaneous cytologic examination or biopsy, bronchoscopy, surgical procedure mediastinoscopy/otmy, and thorascopy/otmy.
Cancer yield rate | Through completion of follow-up (estimated to be 1 year)
Adverse event rate for screening | Through completion of follow-up (estimated to be 1 year)
Number of women with varying Stage (1-4) findings in the lung screening radiology report. | Through completion of follow-up (estimated to be 1 year)
  Histologic type (Bronchioloalveolar carcinoma, adenocarcinoma, squamous-cell carcinoma, large-cell carcinoma, non-small-cell carcinoma or other, small-cell carcinoma, carcinoid).
Cause of death | Through completion of follow-up (estimated to be 1 year)
  Neoplasm of bronchus and lung, other neoplasm, cardiovascular illness, respiratory illness, complications of medical or surgical care, other.

CONTACTS AND LOCATIONS:
Overall Officials: Beryne Odeny, M.D., MPH, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital West County, Creve Coeur, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share results interpretations.
Supporting Information: Study Protocol, SAP
Time Frame: For a period of 1 year.
Access Criteria: Contact the Principal Investigator or Central Contact Back-up via email.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu